CLINICAL TRIAL: NCT05365581
Title: A Phase 1/1b Study of ASP2138 as Monotherapy and in Combination With Pembrolizumab and mFOLFOX6 or Ramucirumab and Paclitaxel in Participants With Metastatic or Locally Advanced Unresectable Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma and in Combination With mFOLFIRINOX in Participants With Metastatic or Locally Advanced Unresectable Pancreatic Adenocarcinoma Whose Tumors Have Claudin (CLDN) 18.2 Expression
Brief Title: A Study of ASP2138 Given by Itself or Given With Other Cancer Treatments in Adults With Stomach Cancer, Gastroesophageal Junction Cancer, or Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2138-CL-0101; jRCT2031210644 (Registry Identifier: jRCT); CTR20241945 (Registry Identifier: chinadrugtrials.org.cn); 2023-504514-29 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-05-05; First posted 2022-05-09 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction (GEJ) Adenocarcinoma; Pancreatic Adenocarcinoma
Keywords: Claudin (CLDN) 18.2; ASP2138; Pharmacokinetics; Safety; Tolerability
MeSH Terms: conditions — Adenocarcinoma | interventions — pembrolizumab; Oxaliplatin; Leucovorin; Fluorouracil; Ramucirumab; Paclitaxel; Irinotecan; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Monotherapy Dose Escalation (Phase 1) (Experimental): A dose escalation design will be used to determine the Maximum Tolerated Dose (MTD) and/ or the Recommended Phase 2 Dose (RP2D) regimens to be further evaluated in the Monotherapy Dose Expansion arms.
  Monotherapy Dose escalation part consists of six parts (Part A, B, C, D, E, and F), and approximately 86 patients would be enrolled in total. Participants will be assigned to sequentially escalating dose cohorts of ASP2138 in each part. The study will open with the Part A dosing schedule, while subsequent cohorts will be opened sequentially or in parallel based upon sponsor review of emerging data.
  Interventions: Drug: ASP2138
- Monotherapy Dose Expansion (Phase 1b) Gastric/GEJ cancer (Experimental): Participants will receive ASP2138 at the candidate RP2D regimens determined in Monotherapy Dose Escalation arm.
  Interventions: Drug: ASP2138
- Monotherapy Dose Expansion (Phase 1b) Pancreatic cancer (Experimental): Participants will receive ASP2138 at the candidate RP2D regimens determined in Monotherapy Dose Escalation arm.
  Interventions: Drug: ASP2138
- Combination Therapy Dose Escalation (Phase 1) Part G - First-line Gastric/GEJ Cancer (Experimental): A dose escalation design will be used to determine the MTD and/ or the RP2D regimens to be further evaluated in the Combination Dose Expansion arms.
  In combination dose escalation part G approximately 24 patients would be enrolled in total. Participants will be assigned to sequentially escalating dose cohorts of ASP2138 in combination with pembrolizumab and mFOLFOX6 as first line therapy.
  Interventions: Drug: ASP2138; Drug: Pembrolizumab; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil
- Combination Therapy Dose Escalation (Phase 1) Part H - Second-line Gastric/GEJ Cancer (Experimental): A dose escalation design will be used to determine the MTD and/ or the RP2D regimens to be further evaluated in the Combination Dose Expansion arms.
  Participants will be assigned to sequentially escalating dose cohorts of ASP2138 in combination with ramucirumab and paclitaxel as second line therapy.
  Interventions: Drug: ASP2138; Drug: Ramucirumab; Drug: Paclitaxel
- Combination Therapy Dose Escalation (Phase 1) Part I - First line Pancreatic Cancer (Experimental): A dose escalation design will be used to determine the MTD and/ or the RP2D regimens to be further evaluated in the Combination Dose Expansion arms.
  Participants will be assigned to sequentially escalating dose cohorts of ASP2138 in combination with mFOLFIRINOX as first line therapy.
  Interventions: Drug: ASP2138; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil; Drug: Irinotecan
- ASP2138 + Pembrolizumab & mFOLFOX6 Combination Therapy Dose Expansion (Phase 1b) Gastric/GEJ Cancer (Experimental): Participants will receive candidate RP2D regimens of ASP2138 in combination with pembrolizumab & mFOLFOX6 as first line therapy determined in Combination Therapy Dose Escalation arm.
  Interventions: Drug: ASP2138; Drug: Pembrolizumab; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil
- ASP2138 + Ramucirumab & Paclitaxel Combination Therapy Dose Expansion (Phase 1b) Gastric/GEJ Cancer (Experimental): Participants will receive candidate RP2D regimens of ASP2138 in combination with ramucirumab and paclitaxel as second line therapy determined in Combination Therapy Dose Escalation arm.
  Interventions: Drug: ASP2138; Drug: Ramucirumab; Drug: Paclitaxel
- ASP2138 + mFOLFIRINOX Combination Therapy Dose Expansion (Phase 1b) Pancreatic Cancer (Experimental): Participants will receive candidate RP2D regimens of ASP2138 in combination with mFOLFIRINOX as first line therapy in pancreatic cancer determined in Combination Therapy Dose Escalation arm in combination with mFOLFIRINOX as first line therapy in pancreatic cancer.
  Interventions: Drug: ASP2138; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil; Drug: Irinotecan
- ASP2138 + Pembrolizumab & CAPOX CTDE Exploratory Cohort (Phase1b) Gastric/GEJ Cancer - Japan & Korea (Experimental): Participants will receive candidate RP2D regimens of ASP2138 in combination with pembrolizumab & CAPOX as first line therapy determined in Combination Therapy Dose Escalation arm.
  CTDE: Combination Therapy Dose Expansion
  Interventions: Drug: ASP2138; Drug: Pembrolizumab; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: ASP2138 — Intravenously or Subcutaneously
Drug: Pembrolizumab — Intravenously
  Arms: ASP2138 + Pembrolizumab & CAPOX CTDE Exploratory Cohort (Phase1b) Gastric/GEJ Cancer - Japan & Korea; ASP2138 + Pembrolizumab & mFOLFOX6 Combination Therapy Dose Expansion (Phase 1b) Gastric/GEJ Cancer; Combination Therapy Dose Escalation (Phase 1) Part G - First-line Gastric/GEJ Cancer
Drug: Oxaliplatin — Intravenously
  Arms: ASP2138 + Pembrolizumab & CAPOX CTDE Exploratory Cohort (Phase1b) Gastric/GEJ Cancer - Japan & Korea; ASP2138 + Pembrolizumab & mFOLFOX6 Combination Therapy Dose Expansion (Phase 1b) Gastric/GEJ Cancer; ASP2138 + mFOLFIRINOX Combination Therapy Dose Expansion (Phase 1b) Pancreatic Cancer; Combination Therapy Dose Escalation (Phase 1) Part G - First-line Gastric/GEJ Cancer; Combination Therapy Dose Escalation (Phase 1) Part I - First line Pancreatic Cancer
Drug: Leucovorin — Intravenously
  Other Names: Folinic acid
  Arms: ASP2138 + Pembrolizumab & mFOLFOX6 Combination Therapy Dose Expansion (Phase 1b) Gastric/GEJ Cancer; ASP2138 + mFOLFIRINOX Combination Therapy Dose Expansion (Phase 1b) Pancreatic Cancer; Combination Therapy Dose Escalation (Phase 1) Part G - First-line Gastric/GEJ Cancer; Combination Therapy Dose Escalation (Phase 1) Part I - First line Pancreatic Cancer
Drug: Fluorouracil — Intravenously
  Arms: ASP2138 + Pembrolizumab & mFOLFOX6 Combination Therapy Dose Expansion (Phase 1b) Gastric/GEJ Cancer; ASP2138 + mFOLFIRINOX Combination Therapy Dose Expansion (Phase 1b) Pancreatic Cancer; Combination Therapy Dose Escalation (Phase 1) Part G - First-line Gastric/GEJ Cancer; Combination Therapy Dose Escalation (Phase 1) Part I - First line Pancreatic Cancer
Drug: Ramucirumab — Intravenously
  Arms: ASP2138 + Ramucirumab & Paclitaxel Combination Therapy Dose Expansion (Phase 1b) Gastric/GEJ Cancer; Combination Therapy Dose Escalation (Phase 1) Part H - Second-line Gastric/GEJ Cancer
Drug: Paclitaxel — Intravenously
  Arms: ASP2138 + Ramucirumab & Paclitaxel Combination Therapy Dose Expansion (Phase 1b) Gastric/GEJ Cancer; Combination Therapy Dose Escalation (Phase 1) Part H - Second-line Gastric/GEJ Cancer
Drug: Irinotecan — Intravenously
  Arms: ASP2138 + mFOLFIRINOX Combination Therapy Dose Expansion (Phase 1b) Pancreatic Cancer; Combination Therapy Dose Escalation (Phase 1) Part I - First line Pancreatic Cancer
Drug: Capecitabine — Oral Administration
  Arms: ASP2138 + Pembrolizumab & CAPOX CTDE Exploratory Cohort (Phase1b) Gastric/GEJ Cancer - Japan & Korea

SUMMARY:
Claudin 18.2 protein, or CLDN18.2 is a protein found on cells in the digestive system. It is also found on some tumors. Researchers are looking at ways to attack CLDN18.2 to help control tumors. ASP2138 is thought to bind to CLDN18.2 and a protein on a type of immune cell called a T-cell. This "tells" the immune system to attack the tumor. ASP2138 is a potential treatment for people with stomach cancer, gastroesophageal junction cancer (GEJ cancer) or pancreatic cancer. GEJ is where the tube that carries food (esophagus) joins the stomach. Before ASP2138 is available as a treatment, the researchers need to understand how it is processed by and acts upon the body. In this study, ASP2138 will either be given by itself, or given together with standard treatments for gastric, GEJ and pancreatic cancer. Pembrolizumab and mFOLFOX6, and ramucirumab and paclitaxel are standard treatments for gastric and GEJ cancer. mFOLFIRINOX is a standard treatment for pancreatic cancer. This information will help find a suitable dose of ASP2138 given by itself and together with the standard cancer treatments and to check for potential medical problems from the treatments.

The main aims of the study are:

* To check the safety of ASP2138 and how well people can tolerate medical problems during the study.
* To find a suitable dose of ASP2138 to be used later in the study.
* These are done for ASP2138 given by itself and when given together with the standard cancer treatments.

Adults 18 years or older with stomach cancer, GEJ cancer, or pancreatic cancer can take part. Their cancer is locally advanced unresectable or metastatic. Locally advanced means the cancer has spread to nearby tissue. Unresectable means the cancer cannot be removed by surgery. Metastatic means the cancer has spread to other parts of the body. There should also be the CLDN18.2 marker in a tumor sample. People cannot take part if they need to take medicines to suppress their immune system, have blockages or bleeding in their gut, have specific uncontrollable cancers, have specific infections, have a condition such as hemophagocytic lymphohistiocytosis (HLH) which is when the body over-reacts to a "trigger" such as infection, or have a specific heart condition ("New York Heart Association Class III or IV").

Phase 1: Lower to higher doses of ASP2138

* ASP2138 is either given through a vein (intravenous infusion) or just under the skin (subcutaneous injection).
* Different small groups are given lower to higher doses of ASAP2138.
* ASP2138 is either given by itself, or given with 1 of 3 standard treatments:
* Pembrolizumab and mFOLFOX6 (first treatment for gastric GEJ cancer)
* Ramacirumab and paclitaxel (Second treatment for gastric or GEJ cancer)
* ASP2138 with mFOLFIRINOX (first treatment for pancreatic cancer)

Phase 1b: doses of ASP2138 worked out from Phase 1

* ASP2138 is either given through a vein or just under the skin. This depends on the findings from Phase 1.
* People with gastric cancer, GEJ cancer or pancreatic cancer are given doses of ASP2138, worked out from Phase 1.
* This includes doses of ASP2138 given by itself and ASP2138 given with the standard cancer treatments.
* The standard cancer treatments given depends on the type of cancer they have.

End of treatment visit: This is 7 days after final dose of study treatment or if the study doctor decides to stop the person's treatment.

People who have locally advanced unresectable pancreatic cancer will not receive ASP2138 by itself.

ELIGIBILITY:
Inclusion Criteria:

* Participant is considered an adult according to local regulation at the time of signing the informed consent form (ICF).
* Female participant is not pregnant, confirmed by serum pregnancy test &vmedical evaluation by interview & at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 6 months after final study intervention administration.
* Female participant must agree not to breastfeed starting at screening & throughout the study period & for 6 months after the final study intervention administration.
* Female participant must not donate ova starting at screening & throughout the study period & for 6 months after the final study intervention administration.
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period & for 6 months after the final study intervention administration.
* Male participant must not donate sperm during the treatment period & for 6 months after the final study intervention administration.
* Male participant with pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study period & for 6 months after the final study intervention administration.
* Participant's tumor sample is positive for claudin (CLDN)18.2 expression by central immunohistochemistry (IHC) testing.
* Participant has radiographically-confirmed, locally advanced, unresectable or metastatic disease within 28 days prior to the first dose of study intervention.
* Participant has at least 1 measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 within 28 days prior to the first dose of study intervention. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Participant has QT interval by Fredericia (QTcF) =< 470 msec.
* Participant agrees not to participate in another interventional study while receiving study Intervention in the present study.
* Participant has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participant has predicted life expectancy >= 12 weeks.
* Participant must meet all of criteria based on laboratory tests within 7 days prior to the first dose of study Intervention. In case of multiple laboratory data within this period, the most recent data should be used. If a participant has received a recent blood transfusion, the laboratory tests must be obtained >= 1 week after any blood transfusion.

Monotherapy Disease specific Criteria: Gastric/GEJ Cancer

* Participant has histologically confirmed metastatic, locally advanced unresectable gastric/gastroesophageal junction (GEJ) adenocarcinoma.
* Escalation: Participant with gastric/GEJ adenocarcinoma who has progressed, is intolerant, has refused, or for whom there is no standard approved therapies that impart significant clinical benefit (no limit to the number of prior treatment regimens).

  * Unique to South Korea: Participant with gastric/GEJ adenocarcinoma who has refused standard approved therapies is not allowed.
* Expansion: Participant with gastric/GEJ adenocarcinoma must have received no more than 3 prior lines of systemic chemotherapy treatment.

  * Unique to EU: Expansion: Participant with gastric/GEJ adenocarcinoma must have received at least first-line standard therapies in the metastatic setting, must have received ramucirumab treatment if eligible & where ramucirumab is available, & no more than 3 prior lines of systemic chemotherapy treatment.

Monotherapy Disease specific Criteria: Pancreatic Cancer

* Participant has histologically or cytologically confirmed metastatic pancreatic adenocarcinoma.
* Escalation: Participant with pancreatic adenocarcinoma who has progressed, is intolerant, has refused, or for whom there is no standard approved therapies that impart significant clinical benefit (no limit to the number of prior treatment regimens).

  * Unique to South Korea: Participant with pancreatic adenocarcinoma who has refused standard approved therapies is not allowed.
* Expansion: Participants with pancreatic adenocarcinoma must have received no more than 2 prior lines of systemic chemotherapy treatment.

Note: Participants with locally advanced unresectable pancreatic adenocarcinoma will not be admitted in monotherapy arms.

* Unique to EU: Participant with pancreatic adenocarcinoma must have received at least first-line standard therapies in the metastatic setting & no more than 2 prior lines of systemic chemotherapy treatment.

For all participants in combination therapy (CT) administration:

* If a participant has received a recent blood transfusion, the laboratory tests must be obtained ≥ 1 week after any blood transfusion.

Combination Therapy Disease-specific (CTDS) Inclusion Criteria: ASP2138 in Combination with Pembrolizumab & mFOLFOX6 as First-line Therapy in Gastric/GEJ Cancer

* Participant has histologically confirmed diagnosis of gastric/GEJ adenocarcinoma.
* Participant has metastatic or locally advanced unresectable gastric/GEJ adenocarcinoma.
* Participant with gastric/GEJ adenocarcinoma has progressed & must not have been previously treated for metastatic disease with either chemotherapy or prior checkpoint inhibitor therapy.
* Participant has a human epidermal growth factor receptor 2 (HER2)-negative tumor per local testing.
* For CT with oxaliplatin, follow contraception guidelines from time of informed consent through at least 9 months after final study intervention.

(Unique to South Korea: For CT with oxaliplatin, follow contraception guidelines from time of informed consent through at least 15 months after final study intervention for women & 12 months after final study intervention for men).

Unique to EU:

* Participant must have a PD-L1 CPS ≥ 1.

CTDS Inclusion Criteria: ASP2138 in Combination with Ramucirumab & Paclitaxel as Second-line Therapy in Gastric/GEJ Cancer

* Participant has histologically confirmed diagnosis of gastric/GEJ adenocarcinoma.
* Participant has metastatic or locally advanced unresectable gastric/GEJ adenocarcinoma.
* Participant with gastric/GEJ adenocarcinoma must have previously received 1 line of systemic chemotherapy treatment (i.e., documented objective radiological or clinical disease progression after first line platinum & fluoropyrimidine treatment in the metastatic setting or disease progression during or within 4 months of the last dose of perioperative treatment.

CTDS Inclusion Criteria: ASP2138 in Combination with mFOLFIRINOX as First-line Therapy in Pancreatic Cancer

* Participant has histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma.
* Participant has confirmed metastatic or locally advanced unresectable pancreatic adenocarcinoma.
* Participant has pancreatic adenocarcinoma, has progressed & must not have received prior systemic anticancer therapy for their advanced disease.
* For CT with oxaliplatin, follow contraception guidelines from time of informed consent through at least 9 months after final study intervention.

(Unique to South Korea: For CT with oxaliplatin, follow contraception guidelines from time of informed consent through at least 15 months after final study intervention for women & 12 months after final study intervention for men).

Japan & Korea Specific:

For All Participants in ASP2138 in Combination with Pembrolizumab & CAPOX:

- If a participant has received a recent blood transfusion, the laboratory tests must be obtained ≥ 1 week after any blood transfusion.

CTDS Inclusion Criteria: ASP2138 in Combination with Pembrolizumab & CAPOX as First-line Therapy in Gastric/GEJ Cancer

* Participant has histologically confirmed diagnosis of gastric/GEJ adenocarcinoma.
* Participant has metastatic or locally advanced unresectable gastric/GEJ adenocarcinoma.
* Participant with gastric/GEJ adenocarcinoma must not have been previously treated for metastatic disease with either chemotherapy or prior checkpoint inhibitor therapy.
* Participants have a HER2-negative tumor per local testing.
* For CT with oxaliplatin, follow contraception guidelines from time of informed consent through at least 9 months after final study intervention.

Exclusion Criteria:

* Participant has received other investigational agents, or antineoplastic therapy including other immunotherapy or devices concurrently or within 21 days or 5 times the half-life, whichever is shorter, prior to first dose of study intervention administration.
* Participant has any condition which makes the participant unsuitable for study participation.
* Participant has known immediate or delayed hypersensitivity or contraindication to any component of study intervention.
* Participant has had prior severe allergic reaction or intolerance to known ingredients of ASP2138 or other antibodies, including humanized or chimeric antibodies.
* Participant weighs < 40 kg.
* Participant has received systemic immunosuppressive therapy, including systemic corticosteroids 14 days prior to first dose of study intervention. Participant using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 10 mg per day of prednisone or equivalent), receiving a single daily dose of systemic corticosteroids or receiving systemic corticosteroids as pre-medication for radiologic imaging contrast use are allowed.
* Participant has a complete gastric outlet syndrome or a partial gastric outlet syndrome with persistent/recurrent vomiting.
* Participant has significant gastric bleeding &/or untreated gastric ulcers that exclude the participant from participation.
* Participant has symptomatic CNS metastases or participant has evidence of unstable CNS metastases even if asymptomatic (e.g., progression on scans). Participants with previously treated CNS metastases are eligible, if they are clinically stable & have no evidence of CNS progression by imaging for at least 4 weeks prior to start of study intervention & are not requiring immunosuppressive doses of systemic steroids (> 10 mg per day of prednisone or equivalent) for longer than 2 weeks.
* Participant is known to have HIV infection. However, participants with cluster of differentiation (CD4) + T cell counts >= 350 cells/µL & no history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections within the past 6 months are eligible. NOTE: Screening for human immunodeficiency virus (HIV) infection should be conducted per local requirements.
* Participant is known to have active hepatitis B (positive hepatitis B surface antigen [HBsAg]) or hepatitis C infection. Testing is required for known history of these infections or as mandated by local requirements. NOTE: Screening for these infections should be conducted per local requirements.

  * For participant who is negative for HBsAg, but hepatitis B core antibody (HBc Ab) positive, a hepatitis B virus (HBV) deoxyribonucleic acid (DNA) test will be performed & if positive the participant will be excluded.
  * Participant with positive hepatitis C virus (HCV) serology, but negative HCV ribonucleic acid (RNA) test results are eligible.
  * Participant treated for HCV with undetectable viral load results are eligible
* Participant has had within 6 months prior to first dose of study intervention any of the following: unstable angina, myocardial infarction, ventricular arrhythmia requiring intervention or hospitalization for heart failure.
* Participant has active infection requiring systemic therapy that has not completely resolved within 7 days prior to the start of study intervention.
* Participant has active autoimmune disease that has required systemic immunosuppressive treatment within the past 1 month prior to the start of study intervention.
* Participant has a clinically significant disease or co-morbidity that may adversely affect the safe delivery of treatment within this study or make the participant unsuitable for study participation.
* Participant has psychiatric illness or social situations that would preclude study compliance.
* Participant has had a major surgical procedure 28 days before start of study intervention & has not fully recovered.
* Participant has received radiotherapy metastatic or for locally advanced unresectable gastric/GEJ or metastatic pancreatic adenocarcinoma 14 days prior to start of study intervention & has NOT recovered from any related toxicity.
* Participant has another malignancy for which treatment is required.
* Participant who has received CLDN18.2-targeted therapy (e.g., zolbetuximab or chimeric antigen receptor CLDN18.2-specific T cells) prior to first dose of study intervention administration is not eligible for dose escalation cohorts. However, a participant who has received CLDN18.2-targeted therapy greater than 28 days or 5 half-lives (whichever is longer) prior to first dose study intervention administration is eligible for dose expansion cohorts only, with the exception of participants who have experienced Grade >= 3 gastrointestinal toxicity after receiving an CLDN18.2-targeted therapy.
* Participant has a history or complication of interstitial lung disease.

China Specific:

Participant who has received treatment with herbal medications that have known antitumor activity within 28 days prior to first dose of study treatment.

For all participants in CT administration:

* Participant has prior severe allergic reaction; suspected, known immediate or delayed hypersensitivity; or intolerance or contraindication to any study intervention (i.e., pembrolizumab & mFOLFOX6 [all components], ramucirumab & paclitaxel or mFOLFIRINOX [all components]).
* For 5 FU (fluorouracil): Participant has known dihydropyrimidine dehydrogenase (DPD) deficiency. (NOTE: Screening for DPD deficiency should be conducted per local requirements).
* Participants who have received systemic immunosuppressive therapy, including systemic corticosteroids 14 days prior to the first dose of study intervention are generally excluded; however, participants using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 10 mg per day of prednisone or equivalent), receiving a single daily dose of systemic corticosteroids or receiving systemic corticosteroids as pre-medication for radiologic imaging contrast or for chemotherapy (as part of CT administration) are allowed.
* Participant is known to have HIV infection.
* NOTE: Differing from monotherapy administration, participants with CD4+ T cell counts ≥ 350 cells/µL & no history of AIDS-defining opportunistic infections within the past 6 months remain ineligible.
* NOTE: Screening for HIV infection should be conducted per local requirements.
* Participant has had uncontrolled high blood pressure within 6 months prior to the first dose of study intervention (Unique to EU: high blood pressure Stage 2 is defined as ≥ 140/90 mmHg).
* Participant has a history of ascites requiring drainage more than twice in the past 7 days.

CTDS Exclusion Criteria: ASP2138 in Combination with Pembrolizumab & mFOLFOX6 as First-line Therapy in Gastric/GEJ Cancer:

* Participant has history of (non-infectious) pneumonitis that required steroids, current pneumonitis, or has a history of interstitial lung disease.
* Participant received live-virus vaccination within 30 days prior to the first dose of study intervention.
* Participant has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention or has been diagnosed with an autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Patients that require replacement therapy (e.g., thyroxine [T4], insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) may be enrolled.

CTDS Exclusion Criteria: ASP2138 in Combination with Ramucirumab & Paclitaxel as Second-line Therapy in Gastric/GEJ Cancer:

* History of cerebrovascular accident or transient ischemic attack within 6 months prior to study intervention.
* Participant has significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to study intervention.
* Participant has evidence of a bleeding diathesis or significant coagulopathy.
* Participant has initiated new treatment with medications that affect the coagulation cascade with an INR ≥ 2 such as vitamin K antagonists, heparins & direct thrombin inhibitors or the use of factor Xa inhibitors within 28 days prior to the start of study intervention.

Note: If the participant started receiving such medications more than 28 days prior to the start of study intervention & needs to continue, this is allowed. However, new anticoagulation medications may not be initiated within 28 days prior to the start of study intervention.

Japan & Korea Specific:

For All Participants in ASP2138 in Combination with Pembrolizumab & CAPOX:

* Participant has prior severe allergic reaction; suspected, known immediate or delayed hypersensitivity; or intolerance or contraindication to any study intervention (i.e., pembrolizumab & CAPOX [all components]).
* Participants who have received systemic immunosuppressive therapy, including systemic corticosteroids 14 days prior to the first dose of study intervention are generally excluded, however, participants using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 10 mg per day of prednisone or equivalent), receiving a single dose of systemic corticosteroids or receiving systemic corticosteroids as pre-medication for radiologic imaging contrast or for chemotherapy (as part of CT administration) are allowed.
* Participant is known to have HIV infection.
* NOTE: Differing from monotherapy administration, participants with CD4+ T cell counts ≥ 350 cells/μL & no history of AIDS-defining opportunistic infections within the past 6 months remain ineligible.
* NOTE: Screening for HIV infection should be conducted per local requirements.
* Participant has had uncontrolled high blood pressure within 6 months prior to the first dose of study intervention.
* Participant has a history of ascites requiring drainage more than twice in the past 7 days.
* Participant has known DPD deficiency. (NOTE: Screening for DPD deficiency should be conducted per local requirements).

CTDS Exclusion Criteria:

ASP2138 in Combination with Pembrolizumab & CAPOX as First-line Therapy in Gastric/GEJ Cancer:

* Participant has history of (noninfectious) pneumonitis that required steroids, current pneumonitis, or has a history of interstitial lung disease.
* Participant received live-virus vaccination within 30 days prior to the first dose of study intervention.
* Participant has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention or has been diagnosed with an autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Participants who require replacement therapy (e.g., thyroxine [T4], insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) may be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) (Phase 1 Dose Escalation) | Up to 28 days
  A DLT is defined as any of the prespecified Adverse Events (AEs) (graded using National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE] version 5.0, except cytokine release syndrome [CRS] and immune effector cell-associated neurotoxicity syndrome [ICANS] which are graded using American Society for Transplantation and Cellular Therapy [ASTCT] consensus grading) or laboratory findings that the investigator or sponsor cannot clearly attribute to a cause other than study drug occurring during the DLT evaluation period.
Number of participants with Adverse Events (AEs) | Up to 27 months
  An AE is any untoward medical occurrence temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. This includes events related to the comparator and events related to the (study) procedures.
Number of participants with serious AEs (SAEs) | Up to 27 months
  An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or other medically important events.
Number of participants with laboratory value abnormalities | Up to 25 months
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities | Up to 27 months
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiogram (ECG) abnormalities | Up to 24 months
  Number of participants with potentially clinically significant ECG values.
Number of participants with physical exam abnormalities | Up to 25 months
  Number of participants with potentially clinically significant physical exam values.
Number of participants at each grade of the Eastern Cooperative Oncology Group (ECOG) performance status | Up to 25 months
  The ECOG scale will be used to assess performance status. Grades range from 0 (fully active) to 5 (dead). Negative change scores indicate an improvement. Positive scores indicate a decline in performance.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ASP2138 in serum: Area under the concentration-time curve (AUC) from the time of dosing to the start of the next dosing interval at multiple dose conditions (AUCtau) | Up to 12 months
  AUCtau will be recorded from the PK serum samples collected.
PK of ASP2138 in serum: maximum concentration (Cmax) | Up to 12 months
  Cmax will be recorded from the PK serum samples collected.
PK of ASP2138 in serum: concentration immediately prior to dosing at multiple dosing (Ctrough) | Up to 12 motnhs
  Ctrough will be recorded from the PK serum samples collected.
PK of ASP2138 in serum: time of the maximum concentration (Tmax) | Up to 12 months
  Tmax will be recorded from the PK serum samples collected.
Overall response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (Phase 1b dose expansion) | Up to 21 months
  ORR is defined as the proportion of participants for each dosing scheme whose best overall response is rated as confirmed complete response (CR) or partial response (PR) per RECIST 1.1.
Disease control rate (DCR) per RECIST 1.1 (Phase 1b dose expansion) | Up to 21 months
  DCR is defined as the proportion of participants for each dosing scheme whose best overall response is rated as confirmed CR, PR or stable disease (SD) per RECIST 1.1.
Change from baseline in serum carbohydrate antigen 19-9 (CA19-9) (pancreatic only) (Phase 1b dose expansion) | up to 21 months
  Serum CA19-9 level will be assessed by local laboratory in participants with pancreatic cancer.
Change from baseline in claudin (CLDN) 18.2 tumor expression level | Up to 6 weeks
  Comparison of CLDN18.2 expression in baseline versus on-treatment tumor biopsies will be performed.
Change from baseline in programmed death-ligand 1 (PD-L1) tumor expression level | Up to 6 weeks
  Comparison of PD-L1 expression in baseline versus on-treatment tumor biopsies will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (44):
- United States (13):
  - University of California Irvine Medical Center, Orange, California
  - UCLA Dept of Medicine - Hematology/Oncology, Santa Monica, Santa Monica, California
  - Northwestern University, Chicago, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYU Langone Medical Center - NYU Medical Oncology Associates, New York, New York
  - Columbia University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Children's Hospital and Health Center, Durham, North Carolina
  - Wake Forest University Baptist Health, Winston-Salem, North Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- China (5):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
- France (6):
  - Site FR33005, Vaillant, Villejuif
  - Site FR33003, Lyon
  - Site FR33004, Marseille
  - Site FR33006, Poitiers
  - Site FR33001, Saint-Herblain
  - Site FR33002, Toulouse
- Italy (4):
  - Site IT39004, Milan
  - Site IT39001, Milan
  - Site IT39005, Rozzano
  - Site IT39003, Verona
- Japan (7):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Kindai University Hospital, Sakai, Osaka
  - The University of Osaka Hospital, Suita, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
- Site PR16101, San Juan, Puerto Rico
- South Korea (5):
  - Site KR82004, Seongnam-si, Gyeonggi-do
  - Site KR82001, Guro-gu, Seoul
  - Site KR82002, Jongno-gu, Seoul
  - Site KR82003, Seocho-gu, Seoul
  - Site KR82005, Seodaemun-gu, Seoul
- Spain (3):
  - Site ES34001, Barcelona
  - Site ES34002, Barcelona
  - Site ES34007, El Palmar

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/